CLINICAL TRIAL: NCT03173456
Title: Comparing the Efficacy of Five Oral Analgesics for Treatment of Acute Musculoskeletal Extremity Pain in the Emergency Department
Brief Title: Comparing Five Oral Analgesics for Treatment of Acute Pain in the Emergency Department (ED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Polly Bijur, Professor of Emergency Medicine, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-7322
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Musculoskeletal Pain
Keywords: acute pain; musculoskeletal pain; emergency medicine; Emergency Service, Hospital; analgesics; Acetaminophen; Ibuprofen; oxycodone; hydrocodone; codeine; adult
MeSH Terms: conditions — Musculoskeletal Pain; Acute Pain; Emergencies | interventions — oxycodone-acetaminophen; acetaminophen, hydrocodone drug combination; Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A pharmacist working in an area inaccessible to ED staff will ensure blinding of the study by masking the medication and inserting it into identical unmarked gel capsules, filling any void with small amounts of lactose. Randomization will be performed in blocks of 10 determined by a sequence generated at http://www.randomization.com. The pharmacist will make up numbered research packets based on the random allocation list, each with 5 tablets containing the masked investigational medication. Research packets will be removed sequentially by the nurse from the Pyxis automated medical dispensing system and administered to the study patients in the ED.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- oxycodone/acetaminophen (APAP) (Active Comparator): 5 mg oxycodone + 325 mg acetaminophen
  Interventions: Drug: oxycodone/APAP
- hydrocodone/APAP (Active Comparator): 5 mg hydrocodone + 300 mg acetaminophen
  Interventions: Drug: hydrocodone/APAP
- codeine/APAP (Active Comparator): 30 mg codeine + 300 mg acetaminophen
  Interventions: Drug: codeine/APAP
- 400 ibuprofen/APAP (Active Comparator): 400 mg ibuprofen + 1000 mg acetaminophen
  Interventions: Drug: 400 ibuprofen/APAP
- 800 ibuprofen/APAP (Active Comparator): 800 mg ibuprofen + 1000 mg acetaminophen
  Interventions: Drug: 800 ibuprofen/APAP

INTERVENTIONS:
Drug: oxycodone/APAP — Oxycodone/acetaminophen 5 mg-325 mg oral tablet
  Other Names: Percocet
  Arms: oxycodone/acetaminophen (APAP)
Drug: hydrocodone/APAP — Hydrocodone/Acetaminophen 5 Mg-300 Mg oral tablet
  Other Names: Vicodin
  Arms: hydrocodone/APAP
Drug: codeine/APAP — Codeine/acetaminophen 30 mg-300mg oral tablet
  Other Names: Tylenol # 3
  Arms: codeine/APAP
Drug: 400 ibuprofen/APAP — ibuprofen/acetaminophen 400 mg-1000mg oral tablet
  Other Names: Motrin, Tylenol
  Arms: 400 ibuprofen/APAP
Drug: 800 ibuprofen/APAP — ibuprofen/acetaminophen 800 mg-1000 mg oral tablet
  Other Names: Motrin, Tylenol
  Arms: 800 ibuprofen/APAP

SUMMARY:
This study compares the efficacy of five oral analgesics: 5 mg oxycodone + 325 mg acetaminophen, 5 mg hydrocodone + 300 mg acetaminophen, 30 mg codeine + 300 mg acetaminophen, 400 mg ibuprofen + 1000 mg acetaminophen, and 800 mg ibuprofen + 1000 mg acetaminophen for the treatment of patients with acute musculoskeletal pain who present to the Emergency Department (ED).

DETAILED DESCRIPTION:
The optimal treatment of musculoskeletal extremity pain in the ED not known. The study is a randomized controlled trial designed to compare the efficacy of five oral analgesics: 5 mg oxycodone + 325 mg acetaminophen, 5 mg hydrocodone + 300 mg acetaminophen, 30 mg codeine + 300 mg acetaminophen, 400 mg ibuprofen + 1000 mg acetaminophen, and 800 mg ibuprofen + 1000 mg acetaminophen for the treatment of patients with acute musculoskeletal pain. The primary outcome is the between treatment group difference in change in patients' rating of pain intensity one hour after ingestion of the study medication. Secondary outcomes include: 1) the between treatment group difference in change in patients' rating of pain intensity two hours after ingestion of the study medication; 2) difference in proportion of patients who receive rescue medication; 3) difference in proportion of patients who would choose to take the study medication again if they returned to the ED with similar pain; 4) difference in proportion of patients who experience side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 21 through 64 years of age
* Complaint of acute musculoskeletal pain in one or more extremity, defined as distal to and including the shoulder or hip joints.
* Pain of less than seven days duration
* Patient speaks Spanish or English
* The clinician plans to treat the patient in the ED with oral analgesics and is willing to treat the patient with opioid analgesics or up to 800 mg ibuprofen and 1000 mg acetaminophen
* Patient is going to receive imaging of the painful extremity
* Clinician judges patient to have capacity to provide informed consent

Exclusion Criteria:

* Patient does not have cell phone or cannot receive a verification phone call on their cell phone while in the ED
* Any use of methadone currently or previously
* Chronic condition requiring frequent pain management such as arthritis, sickle cell disease, fibromyalgia, or any neuropathy
* History of an adverse reaction to any of the study medications
* Opioids taken in the past 24 hours
* Ibuprofen or acetaminophen taken in past 24 hours
* Any other prescribed or over the counter topical or oral analgesics taken in past 24 hrs
* Pregnancy by either urine or serum human chorionic gonadotropin testing
* Breastfeeding per patient report
* History of peptic ulcer disease
* Medical condition that might affect metabolism of opioid analgesics, acetaminophen, or ibuprofen such as hepatitis, renal insufficiency, hypo- or hyperthyroidism, Addison's, or Cushing's disease
* Lacerations,
* Multiple injuries
* Taking any medicine that might interact with one of the study medications, such as antidepressant SSRI's or tricyclics, antipsychotics, anti-malaria medications quinidine or halofantrine, amiodarone or dronedarone, diphenhydramine, celecoxib, ranitidine, cimetidine, ritonavir, terbinafine, or St John's Wort

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Friedman, MD, Study Director — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bijur PE, Friedman BW, Irizarry E, Chang AK, Gallagher EJ. A Randomized Trial Comparing the Efficacy of Five Oral Analgesics for Treatment of Acute Musculoskeletal Extremity Pain in the Emergency Department. Ann Emerg Med. 2021 Mar;77(3):345-356. doi: 10.1016/j.annemergmed.2020.10.004. Epub 2020 Dec 23. PMID 33358232

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited when they came into the ED with a complaint of pain. They were recruited in 2 academic EDs by trained, full-time, bilingual research associates from 11/26/2017 to 11/5/2019
Period: Baseline
Arm/Group | Oxycodone/Acetaminophen (APAP) | Hydrocodone/APAP | Codeine/APAP | 400 Ibuprofen/APAP | 800 Ibuprofen/APAP
Started | 120 | 120 | 120 | 120 | 120
Completed | 120 | 119 | 120 | 120 | 118
Not Completed | 0 | 1 | 0 | 0 | 2
Not completed — Medication dispensing system malfunction' | 0 | 1 | 0 | 0 | 2
Period: 2 Hour Follow-up
Arm/Group | Oxycodone/Acetaminophen (APAP) | Hydrocodone/APAP | Codeine/APAP | 400 Ibuprofen/APAP | 800 Ibuprofen/APAP
Started | 120 | 119 | 120 | 120 | 118
Completed | 120 | 118 | 119 | 119 | 116
Not Completed | 0 | 1 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The 3 patients assigned to treatment arms did not provide any data because of malfunctioning of the medication dispensing system.
Groups:
- Oxycodone/APAP: 5 mg oxycodone + 325 mg acetaminophen
  oxycodone/APAP: Oxycodone/acetaminophen 5 mg-325 mg oral tablet
- Total: Total of all reporting groups
Arm/Group | Oxycodone/APAP | Hydrocodone/APAP | Codeine/APAP | 400 Ibuprofen/APAP | 800 Ibuprofen/APAP | Total
Number analyzed (Participants) | 120 | 119 | 120 | 120 | 118 | 597
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (12) | 39 (12) | 38 (12) | 36 (12) | 38 (13) | 37.4 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 50 | 59 | 53 | 50 | 265
  Male | 67 | 69 | 61 | 67 | 68 | 332
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 82 | 83 | 32 | 37 | 313
  Not Hispanic or Latino | 40 | 36 | 37 | 87 | 81 | 281
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 4 | 5 | 1 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 47 | 43 | 46 | 32 | 47 | 215
  White | 40 | 37 | 44 | 52 | 46 | 219
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 30 | 36 | 26 | 31 | 24 | 147
Region of Enrollment [Number; unit: participants]
  United States | 120 | 119 | 120 | 120 | 118 | 597
Initial pain intensity scale [Count of Participants; unit: Participants] — Numerical Rating Scale: Scale ranging from 0 "no pain" to 10 "worst imaginable pain" Patients are asked to give number that best represents their pain
  Participants
    0-6 | 5 | 4 | 1 | 3 | 2 | 15
    7 | 14 | 9 | 8 | 6 | 13 | 50
    8 | 16 | 19 | 26 | 19 | 19 | 99
    9 | 19 | 22 | 17 | 22 | 15 | 95
    10 | 66 | 65 | 68 | 70 | 69 | 338
Diagnosis [Count of Participants; unit: Participants]
  Sprain or Strain | 75 | 78 | 68 | 68 | 82 | 371
  Extremity Fracture | 21 | 11 | 17 | 24 | 14 | 87
  Muscle pain | 12 | 13 | 17 | 13 | 11 | 66
  Contusion | 1 | 10 | 11 | 6 | 6 | 34
  Other | 11 | 7 | 7 | 9 | 5 | 39
Non-Pharmacologic interventions [Count of Participants; unit: Participants]
  0 | 63 | 64 | 64 | 55 | 51 | 297
  greater than or equal to 1 | 57 | 55 | 56 | 65 | 67 | 300

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain From Before Medication Administered (Baseline) to One-hour Post-baseline
Description: Pain intensity measured by 11-point Numerical Rating Scale (NRS) of Pain 0 = no pain 10 = worse possible pain. Change calculated as NRS before medication administered (denoted as baseline) minus NRS 1-hour post-baseline. Higher scores mean more change which is the better outcome.
Time Frame: Prior to Ingestion of study medication to one hour after ingestion of the study medication
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | 400 Ibuprofen/APAP | 800 Ibuprofen/APAP | Codeine/APAP | Hydrocodone/APAP | Oxycodone/APAP
Number analyzed (Participants) | 120 | 118 | 120 | 119 | 120
Units on a scale | 3.0 [2.6 to 3.5] | 3.0 [2.5 to 3.5] | 3.4 [2.9 to 3.9] | 3.1 [2.7 to 3.5] | 3.3 [2.8 to 3.7]
Statistical Analysis 1: Comparison: 400 Ibuprofen/APAP vs 800 Ibuprofen/APAP vs Codeine/APAP vs Hydrocodone/APAP vs Oxycodone/APAP; The null hypothesis is that all means are equal. The alternate hypothesis is that one or more mean is less than or more than another; Test type: Superiority; p = 0.69, ANOVA — A priori threshold for statistical significance was 0.05. The plan was to only do individual comparisons between means if the overall test of the analysis of variance (AVOVA) was statistically significant

2. Secondary Outcome: Change in Pain From Before Medication Administered (Baseline) to Two Hour Post-baseline
Description: Pain intensity measured by 11-point Numerical Rating Scale (NRS) of Pain 0 = no pain 10=worst possible pain. Change is calculated as Numerical Rating Scale before medication is administered (denoted as baseline) minus NRS 2- hours past baseline. Higher numbers indicate better outcomes.
Time Frame: Prior to ingestion of study medication to 2 hours after ingestion of the study medication
Population: Differences between population at 1 hour and 2 hour is due to patients leaving the Emergency Department before 2 hours post-baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 400 Ibuprofen/APAP | 800 Ibuprofen/APAP | Codeine/APAP | Hydrocodone/APAP | Oxycodone/APAP
Number analyzed (Participants) | 119 | 116 | 119 | 117 | 120
units on a scale | 4.3 [3.9 to 4.8] | 4.6 [4.1 to 5.1] | 4.4 [3.9 to 4.9] | 4.5 [4.1 to 5.0] | 4.7 [4.2 to 5.2]
Statistical Analysis 1: Comparison: 400 Ibuprofen/APAP vs 800 Ibuprofen/APAP vs Codeine/APAP vs Hydrocodone/APAP vs Oxycodone/APAP; Test type: Superiority; p = 0.85, ANOVA — Threshold for statistical significance was 0.05. The plan was to only compare means if the overall test of AVOVA was statistically significant

3. Secondary Outcome: Percentage of Patients Who Received Rescue Medication
Description: Number of patients who received additional analgesics divided by total number of patients x 100
Time Frame: Entire two-hour time period
Measure: Count of Participants; unit: Participants
Arm/Group | 400 Ibuprofen/APAP | 800 Ibuprofen/APAP | Codeine/APAP | Hydrocodone/APAP | Oxycodone/APAP
Number analyzed (Participants) | 119 | 116 | 119 | 118 | 120
Participants | 29 | 28 | 26 | 27 | 28
Statistical Analysis 1: Comparison: 400 Ibuprofen/APAP vs 800 Ibuprofen/APAP vs Codeine/APAP vs Hydrocodone/APAP vs Oxycodone/APAP; Test type: Superiority; p = 0.99, Chi-squared — Threshold for statistical significance = 0.05

4. Secondary Outcome: Percentage of Patients Who Would Choose to Take the Study Medication Again if They Returned to the ED With Similar Pain
Description: Number of patients who would choose to take study medication again divided by number of patients x 100. Question asked at end of two-hour time period
Time Frame: End of two-hour time period
Population: Missing data: 1 from codeine/APAP arm, 1 from hydrocodone/APAP arm, 2 from oxycodone/APAP arm
Measure: Count of Participants; unit: Participants
Arm/Group | 400 Ibuprofen/APAP | 800 Ibuprofen/APAP | Codeine/APAP | Hydrocodone/APAP | Oxycodone/APAP
Number analyzed (Participants) | 119 | 116 | 118 | 117 | 118
Participants | 78 | 83 | 75 | 89 | 81

5. Secondary Outcome: Percentage of Patients Who Experience Side Effects Within One Hour of Ingestion of Study Medication
Description: Number of patients who experience side effects within one hour ofr ingestion of study medication divided by total number of patients x 100
Time Frame: From time of ingestion of study medication to one hour later
Measure: Count of Participants; unit: Participants
Arm/Group | 400 Ibuprofen/APAP | 800 Ibuprofen/APAP | Codeine/APAP | Hydrocodone/APAP | Oxycodone/APAP
Number analyzed (Participants) | 120 | 118 | 120 | 119 | 120
Participants | 26 | 37 | 33 | 34 | 37
Statistical Analysis 1: Comparison: 400 Ibuprofen/APAP vs 800 Ibuprofen/APAP vs Codeine/APAP vs Hydrocodone/APAP vs Oxycodone/APAP; Test type: Superiority; p = 0.46, Chi-squared

6. Secondary Outcome: Percentage of Patients Who Experience Side Effects in Two Hours After Ingestion of Study Medication
Description: Number of patients who experience side effects in two hours after ingestion of study medication divided by total number of patients x 100
Time Frame: From time of ingestion of study medication to two hours later
Measure: Count of Participants; unit: Participants
Arm/Group | 400 Ibuprofen/APAP | 800 Ibuprofen/APAP | Codeine/APAP | Hydrocodone/APAP | Oxycodone/APAP
Number analyzed (Participants) | 120 | 118 | 120 | 119 | 120
Participants | 31 | 44 | 40 | 51 | 49
Statistical Analysis 1: Comparison: 400 Ibuprofen/APAP vs 800 Ibuprofen/APAP vs Codeine/APAP vs Hydrocodone/APAP vs Oxycodone/APAP; Test type: Superiority; p = 0.0501, Chi-squared — 0.05 was the a priori threshold for statistical significance

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | 400 Ibuprofen/APAP | 800 Ibuprofen/APAP | Codeine/APAP | Hydrocodone/APAP | Oxycodone/APAP
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/118 | 0/120 | 0/119 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/118 | 0/120 | 0/119 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/118 | 0/120 | 0/119 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT03173456/Prot_SAP_000.pdf